CLINICAL TRIAL: NCT01636271
Title: SB-480848 in Major Adverse Cardiovascular Events - Integrated Phase III Summary of Efficacy and Safety
Brief Title: SB-480848 in Major Adverse Cardiovascular Events - Integrated Summary of Efficacy and Safety From the STABILITY Trial (LPL100601) and the SOLID-TIMI-52 Trial (SB-480848/033)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116740
Record Dates: First submitted 2012-05-31; First posted 2012-07-10 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Heart Disease
Keywords: CV Risk; Cardiovascular Disease; Atherosclerosis; Acute coronary syndrome
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Atherosclerosis; Acute Coronary Syndrome | interventions — darapladib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: subjects from LPL100601: randomized subjects in study LPL100601
  Interventions: Drug: darapladib; Drug: placebo
- Group 2: subjects from SB480848/033: randomized subjects in study SB480848/033
  Interventions: Drug: darapladib; Drug: placebo

INTERVENTIONS:
Drug: darapladib — darapladib enteric coated tablets 160 mg
Drug: placebo — placebo

SUMMARY:
The overall objective of this integrated analysis is to evaluate the clinical safety and efficacy of long-term treatment with darapladib enteric coated tablets, 160mg, as compared to placebo when added to standard of care in subjects with clinical manifestations of cardiovascular disease (chronic coronary heart disease (CHD) and post Acute Coronary Syndrome (ACS)). With respect to efficacy, the key purpose of this integrated analysis is to evaluate the effects of darapladib on the following endpoints: urgent coronary revascularization for myoacrdial ischemia, fatal/non-fatal stroke, time to subsequent Major Adverse Cardiovascular Event (MACE), and heart failure requiring hospitalization. The first occurrent of MACE, Major and total coronary events as well as the individual components of MACE will also be evaluated descriptively.

DETAILED DESCRIPTION:
The objective of the integrated safety analysis is to characterize the safety profile of darapladib in subjects with clinical manifestations of cardiovascular disease (chronic coronary heart disease (CHD) and post Acute Coronary Syndrome (ACS)).

The purpose of the integrated efficacy analysis is to test the effects of darapladib on select endpoints which are not part of the testing hierarchies associated with the individual studies, namely: urgent coronary revascularization for myocardial ischemia, stroke, subsequent MACE, and heart failure requiring hospitalization, For all other endpoints, the intent of the integrated analysis is to provide increased precision of the estimated effects of darapladib.

ELIGIBILITY:
Inclusion Criteria:

* This is an integrated analysis therefore inclusion criteria are not applicable.

Exclusion Criteria:

* This is an integrated analysis therefore exclusion criteria are not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with clinical manifestations of cardiovascular disease (chronic coronary heart disease (CHD) or post Acute Coronary Syndrome (ACS)) randomized into the STABILITY trial (LPL100601) or the SOLID-TIMI 52 trial (SB-480848/033).
Sampling Method: Non-Probability Sample
Enrollment: 28855 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The time to first occurrence of urgent coronary revascularization for myocardial ischemia | visits occur at month 1,3,6, and every 6 months thereafter until 1500 first occurrence MACE events have occurred in each study. It is anticipated that the median follow-up time will be approximately 3 years in each study.
  time to the first occurrence of any urgent coronary revascularization for myocardial ischemia
The time to first occurrence of stroke (fatal/non-fatal) | visits occur at month 1,3,6, and every 6 months thereafter until 1500 first occurrence MACE events have occurred in each study. It is anticipated that the median follow-up time will be approximately 3 years in each study.
  time to the first occurrence of stroke (fatal or non-fatal)
The time to subsequent Major Adverse Cardiovascular Events (MACE) | visits occur at month 1,3,6, and every 6 months thereafter until 1500 first occurrence MACE events have occurred in each study. It is anticipated that the median follow-up time will be approximately 3 years in each study.
  time to subsequent composite of MACE (CV death, non-fatal MI or non-fatal stroke)
The time to first occurrence of heart failure requiring hospitalization | visits occur at month 1,3,6, and every 6 months thereafter until 1500 first occurrence MACE events have occurred in each study. It is anticipated that the median follow-up time will be approximately 3 years in each study.
  time to the first occurrence of heart failure requiring hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline